CLINICAL TRIAL: NCT03040622
Title: The Evaluation of Thrombogenicity in Patients Undergoing WATCHMAN Left Atrial Appendage Closure Trial
Status: Completed | Type: Observational
Sponsor: Inova Health Care Services (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-2583
Record Dates: First submitted 2017-01-04; First posted 2017-02-02 (Estimated); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-10

CONDITIONS: Left Atrial Appendage Closure; WATCHMAN Device Implantation
Keywords: WATCHMAN; Left Atrial Appendage Closure; Thrombosis; Platelet Function
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Watchman Left Atrial Appendage Closure
  Interventions: Device: WATCHMAN Left Atrial Appendage Closure

INTERVENTIONS:
Device: WATCHMAN Left Atrial Appendage Closure — WATCHMAN Left Atrial Appendage Closure

SUMMARY:
This study will evaluate thrombogenicity in patients undergoing left atrial appendage closure using the WATCHMAN device. Parameters of thrombosis and platelet function, as well as other bio-markers, will be measure before, during, and after WATCHMAN implantation at several follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject indicated and scheduled for WATCHMAN device implantation at IHVI (Inova Heart and Vascular Institute)
* Subject may be of either sex and of any race, and must be >18 years of age.
* Subject must be willing and able to give appropriate informed consent.
* The subject is able to read and has signed and dated the informed consent document including authorization permitting release of personal health information approved by the investigator's Institutional Review Board (IRB).

Exclusion Criteria:

* Subjects with contraindications for WATCHMAN device implantation

Intracardiac thrombus is visualized by echocardiographic imaging, An atrial septal defect repair or closure device or a patent foramen ovale repair or closure device is present, The LAA (Left atrial appendage) anatomy will not accommodate a device, Any of the customary contraindications for other percutaneous catheterization procedures (e.g., patient size too small to accommodate TEE - transesophageal echocardiography probe or required catheters) or conditions (e.g., active infection, bleeding disorder) are present, There are contraindications to the use of warfarin, aspirin, or clopidogrel, The patient has a known hypersensitivity to any portion of the device material or the individual components such that the use of the WATCHMAN Device is contraindicated

* Ligated or oversewn left atrium
* Concurrent participation in any investigational study.
* Subject likely to not be available to complete all protocol-required study visits or procedures, to the best of the subject's and investigator's knowledge
* History or evidence of any other clinically significant disorder, condition, or disease other than those outlined above that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects >18 years of age scheduled for left atrial appendage closure procedure with the WATCHMAN device.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

REFERENCES:
- [Derived] Gurbel PA, Bliden K, Sherwood M, Taheri H, Tehrani B, Akbari M, Yazdani S, Asgar JA, Chaudhary R, Tantry US. Development of a routine bedside CYP2C19 genotype assessment program for antiplatelet therapy guidance in a community hospital catheterization laboratory. J Thromb Thrombolysis. 2024 Apr;57(4):566-575. doi: 10.1007/s11239-024-02953-8. Epub 2024 Mar 13. PMID 38480590
- [Derived] Sherwood M, Bliden KP, Ilkhanoff L, Venkataraman G, Strickberger A, Yazdani S, McSwain R, Rashid H, Navarese EP, Plummer T, Batchelor W, Chaudhary R, Tantry US, Gurbel PA. Detailed thrombogenicity phenotyping and 1 year outcomes in patients undergoing WATCHMAN implantation: (TARGET-WATCHMAN) a case-control study. J Thromb Thrombolysis. 2020 Oct;50(3):484-498. doi: 10.1007/s11239-020-02205-5. PMID 32601850

RESULTS

PARTICIPANT FLOW:
Groups:
- Watchman Left Atrial Appendage Closure: Patients implanted with WATCHMAN left atrial appendage closure device in a hospital setting
Period: Overall Study
Arm/Group | Watchman Left Atrial Appendage Closure
Started | 35
Completed | 32
Not Completed | 3
Not completed — unable to implant device | 3

BASELINE CHARACTERISTICS:
Arm/Group | Watchman Left Atrial Appendage Closure
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Thrombin Induced Platelet-fibrin Clot Strength (TIP-FCS) Between Patients With and Without Device Related Thrombosis (DRT) Assessed at 1-year of Watchman Implant
Description: Comparison of thrombin induced platelet-fibrin clot strength (TIP-FCS) as measured using thromboelastography (TEG-6s) between patients with and without device related thrombosis (DRT) assessed by transesophageal echocardiogram after left atrial appendage closure (LAAC) with Watchman device. TIP-FCS >67mm has been associated with increased risk of hypercoagulability.
Time Frame: Assessed at 1 year post implant.
Population: The total group was separated into participants with and without DRT and TIP-FCS was compared between groups.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- With Device Related Thrombosis: Patients with device related thrombosis within 1-year of implant
- Without Device Related Thrombosis: Patients without device related thrombosis within 1-year of implant
Arm/Group | With Device Related Thrombosis | Without Device Related Thrombosis
Number analyzed (Participants) | 3 | 29
mm | 68.0 (1.8) | 62.7 (4.7)
Statistical Analysis 1: Comparison: With Device Related Thrombosis vs Without Device Related Thrombosis; Test type: Other; p = 0.06, ANOVA

2. Secondary Outcome: Comparison of Fibrin Clot Strength (FCS) Between Patients With and Without Device Related Thrombosis (DRT) Assessed at 1-year After Watchman Implant
Description: Comparison of fibrin clot strength (FCS) as measured using thromboelastography (TEG-6s) between patients with and without device related thrombosis (DRT) assessed by transesophageal echocardiogram after left atrial appendage closure (LAAC) with Watchman device. FCS >32mm has been associated with increased risk of thrombosis.
Time Frame: Assessed at 1 year post implant.
Population: The total group was separated into participants with and without DRT and FCS was compared between groups.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | With Device Related Thrombosis | Without Device Related Thrombosis
Number analyzed (Participants) | 3 | 29
mm | 35.6 (6) | 24.4 (6.6)
Statistical Analysis 1: Comparison: With Device Related Thrombosis vs Without Device Related Thrombosis; Test type: Other; p = 0.009, ANOVA

3. Secondary Outcome: Comparison of D-dimer Levels Between Patients With and Without Device Related Thrombosis (DRT) Assessed at 1-year of Watchman Implant
Description: Comparison of D-dimer levels as measured using ACL TOP 300 hemostasis testing system between patients with and without device related thrombosis (DRT) assessed by transesophageal echocardiogram after left atrial appendage closure (LAAC) with Watchman device. D-dimer levels >500ng/ml are associated with thrombo-embolic diseases.
Time Frame: Assessed at 1 year post implant
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | With Device Related Thrombosis | Without Device Related Thrombosis
Number analyzed (Participants) | 3 | 29
ng/ml | 1712 (2330) | 283 (213)
Statistical Analysis 1: Comparison: With Device Related Thrombosis vs Without Device Related Thrombosis; Test type: Other; p = 0.001, ANOVA

4. Secondary Outcome: Number of Participants With Major Adverse Clinical Events (MACE) Post Watchman Implant
Description: Number of participants with MACE [all-cause death, systemic or pulmonary embolism, MI (myocardial ischemia) , TIA (transient ischemic attack) , stroke, DRT, and BARC bleeding (2,3, or 5) ] post Watchman implant..
Time Frame: within 1-year post implant
Measure: Count of Participants; unit: Participants
Groups:
- Major Adverse Clinical Events: MACE within 1-year of Watchman implant
Arm/Group | Major Adverse Clinical Events
Number analyzed (Participants) | 32
Participants
  Device Related Thrombosis | 3
  All-Cause Death | 2
  BARC Bleeding | 4
  Pulmonary Embolism | 1
  TIA | 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: Major adverse clinical outcomes monitored include: all-cause death, embolism (systemic or pulmonary), myocardial infarction, TIA, ischemic or hemorrhagic stroke, device related thrombosis, and major bleeding using the Academic Research Consortium (BARC) definition including BARC type 2, 3 or 5. DRT was defined as the presence of a persistent echogenic mobile mass attached to the WATCHMAN device confirmed by transesophageal echocardiography.
Arm/Group | Watchman Left Atrial Appendage Closure
All-Cause Mortality (participants affected / at risk) | 2/32
Serious Adverse Events (participants affected / at risk) | 17/32
Other Adverse Events (participants affected / at risk) | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Watchman Left Atrial Appendage Closure (N=32)
Device Related Thrombosis (Blood and lymphatic system disorders) | 3 (3)
Major Bleeding (Vascular disorders) | 4 (4) — BARC Bleeding (Type 3A)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
TIA (Nervous system disorders) | 1 (1)
Rehospitalization for atrial fibrillation with rapid ventricular rhythm (Cardiac disorders) | 5 (5)
Rehospitalization for pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rehospitalization-injury from a fall (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03040622/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT03040622/ICF_001.pdf